CLINICAL TRIAL: NCT02457767
Title: Optimization of Waiting - Time in the Anesthesia Admissions Ambulance Department of Anaesthesia and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin by Support of a Mobile Application - a Pilot Study
Brief Title: Optimizing of Waiting - Time in the Anesthesia Admissions Ambulance of the Charité - University Medicine Berlin by Support of a Mobile Application - a Pilot Study
Status: Withdrawn | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: Anaest-App
Record Dates: First submitted 2015-03-20; First posted 2015-05-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Waiting-time in the Anaesthesia Admissions Ambulance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study the investigators measure and optimize the patients waiting time in the preanesthetic assessment by integrating an interactive mobile device. The aim of this study is to observe whether the patients mean waiting-time is reduced by the use of a special mobile application (Anaest-App) and, as a result , raises patient-satisfaction.

DETAILED DESCRIPTION:
3000 patients as well as medical doctors receive tablet-devices. The Software (App) installed on these devices coordinates the virtual waiting numbers assigned to each patient-tablet. The medical doctor can virtually call up the next patient in line for preanesthesiologic assessment. After the examination both medical doctors and patients complete a brief questionaire regarding educational level, usability and overall satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of all ages
* Elective surgical procedure

Exclusion Criteria:

* Language inabilities (German)
* Severe hearing - loss and visual impairment
* In-Patient care > 24 h

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients (aged > 4 years) for elective surgery
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Waiting time in the anesthesia admissions ambulance | Participants will be followed for the duration of ambulation ambulance stay, an expected average of 1 hour
  The waiting time will be measured in hours and minutes

SECONDARY OUTCOMES:
Study patient satisfaction | Participants will be followed for the duration of ambulation ambulance stay, an expected average of 1 hour
  The question "How satisfied is the Patient?" is measured during stay in the anesthesia admissions ambulance.This scale ranges from -3 to +3, contains no "0"(forced-choice).
Medical doctor statisfaction | Participants will be followed for the duration of ambulation ambulance stay, an expected average of 1 day
  The question "How satisfied is the medical doctor?" is measured during stay in the anesthesia admissions ambulance.This scale ranges from -3 to +3, contains no "0"(forced-choice).
Tablet - acceptance by study patients | Participants will be followed for the duration of ambulation ambulance stay, an expected average of 1 hour
  The acceptance is measured by a scale ranges from -3 to +3, contains no "0"(forced-choice).
Tablet - acceptance by medical doctor | Participants will be followed for the duration of ambulation ambulance stay, an expected average of 1 day.
  The acceptance is measured by a scale ranges from -3 to +3, contains no "0"(forced-choice).
Duration of examination time | Participants will be followed for the duration of examinationin the ambulance, an expected average of 1 hour.
  The duration of examination time will be measured in hours and minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine Berlin, Charité - Univeristy Medicine Berlin